CLINICAL TRIAL: NCT05305339
Title: Telocytes in Umbilical Cord of Patients With and Without Pre-eclampsia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hatem Awaga, Lecturer of Obstetrics and Gynecology, Sohag University
Other Study IDs: Soh-Med-21-12-44
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Telocytes in Umbilical Cord of Pregnancies Complicated by Chronic Hypertension, Gestational Hypertension and Preeclampsia
Keywords: Telocytes; Umbilical cord; Preeclampsia
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group A (Control group): Singleton pregnancies undergoing elective pre-labour CS at gestational age (34+0 to 40+0) that are otherwise healthy.
  Interventions: Other: Placental and Umbilical cord biopsy
- Group B (Chronic hypertension): It means systolic blood pressure of 140 mm Hg or more, a diastolic blood pressure of 90 mm Hg or more, or both, that is diagnosed or present before pregnancy or before 20 weeks of gestation on two occasions at least 4 hours apart. Hypertension that is diagnosed for the first-time during pregnancy and that does not resolve in the typical postpartum period also is classified as chronic hypertension
  Interventions: Other: Placental and Umbilical cord biopsy
- Group C (Gestational hypertension): It is usually diagnosed when systolic blood pressure is 140 mm Hg or more or a diastolic blood pressure of 90 mm Hg or more, or both, on two occasions at least 4 hours apart after 20 weeks of gestation, in a woman with a previously normal blood pressure. Gestational hypertension is considered severe when the systolic level reaches 160 mm Hg or the diastolic level reaches 110 mm Hg or both.
  Interventions: Other: Placental and Umbilical cord biopsy
- Group D (Preeclampsia): Women with PE fulfilled the criteria if they had hypertension (> 140/90 mmHg) and proteinuria (> 0.3 gm/day or ≥ +1 by dipstick urine analysis at ≥ 20 weeks of gestation or protein-to-creatinine ratio of 0.30 or more). If no proteinuria, hypertension associated with thrombocytopenia, renal or liver impairment, or pulmonary edema was sufficient to diagnose PE as per ACOG Practice Bulletin No .202
  Interventions: Other: Placental and Umbilical cord biopsy

INTERVENTIONS:
Other: Placental and Umbilical cord biopsy — After delivery of the placenta, two tissue fragments, 1st piece about 1x1 cm from the central zone of the maternal surface of the placenta and 2nd piece about 1 x 1 cm from mid segment of umbilical cord will be cut. Each of both samples will be divided and fixed in either a 10% formalin for light microscopic examination or glutaraldehyde 2.5% for Electron microscopic examination. Paraffin-embedded placental tissue sections (4 μm thick) will be used for histological (stained with hematoxylin and eosin) and immunohistochemical examination using primary antibody markers for telocytes CD117, CD34, vimentin, SMA (smooth muscle actin), and the new telocyte marker TMEM16a (DOG-1).

SUMMARY:
Studying the ultrastructural and immunohistochemical characteristics of Telocytes from umbilical cord vessels wall in PE patients compared to control and its relation to severity of disease whether controlled or uncontrolled.

DETAILED DESCRIPTION:
Patients fulfilling the eligibility criteria of the current research will be approached prior to delivery. The attending physician will explain the nature of the study and all patients will be asked to sign an informed consent.

Routine investigations will be performed to all patients including CBC, liver and renal function and urine analysis in addition to albumin creatinine ratio.

Ultrasound scanning including umbilical doppler indices measurement will be done for all cases before delivery using an HDI ultrasound system (AlbiniouTL Ultrasound, Bothell, WA, USA).

Non stress test is routinely done for all hypertensive patients twice weekly as part of routine work up of such patients in our emergency unit using (CTG machine-NSL BT-350 Bistos) (Korea).

Diagnosis of chronic hypertension, gestational hypertension and preeclampsia

1. preeclampsia: Women with PE fulfilled the criteria if they had hypertension (> 140/90 mmHg) and proteinuria (> 0.3 gm/day or ≥ +1 by dipstick urine analysis at ≥ 20 weeks of gestation or protein-to-creatinine ratio of 0.30 or more). If no proteinuria, hypertension associated with thrombocytopenia, renal or liver impairment, or pulmonary edema was sufficient to diagnose PE as per ACOG Practice Bulletin No .202[6].
2. Gestational hypertension:

   It is usually diagnosed when systolic blood pressure is 140 mm Hg or more or a diastolic blood pressure of 90 mm Hg or more, or both, on two occasions at least 4 hours apart after 20 weeks of gestation, in a woman with a previously normal blood pressure [7]. Gestational hypertension is considered severe when the systolic level reaches 160 mm Hg or the diastolic level reaches 110 mm Hg, or both [6].
3. Chronic hypertension:

It means systolic blood pressure of 140 mm Hg or more, a diastolic blood pressure of 90 mm Hg or more, or both, that is diagnosed or present before pregnancy or before 20 weeks of gestation on two occasions at least 4 hours apart. Hypertension that is diagnosed for the first-time during pregnancy and that does not resolve in the typical postpartum period also is classified as chronic hypertension[8].

Patients are finally classified to PE with severe features, PE without severe features, Gestational hypertension (mild and severe), chronic hypertension and chronic hypertension with superimposed PE and termination will be done according to the recent recommendation of ACOG [6, 8].

Tissue and samples procurement and processing:

Specimen preparation After delivery of the placenta, two tissue fragments, 1st piece about 1x1 cm from the central zone of the maternal surface of the placenta and 2nd piece about 1 x 1 cm from mid segment of umbilical cord will be cut. Each of both samples will be divided and fixed in either a 10% formalin for light microscopic examination or glutaraldehyde 2.5% for Electron microscopic examination. Paraffin-embedded placental tissue sections (4 μm thick) will be used for histological (stained with hematoxylin and eosin) and immunohistochemical examination using primary antibody markers for telocytes CD117, CD34, vimentin, SMA (smooth muscle actin), and the new telocyte marker TMEM16a (DOG-1).

ELIGIBILITY:
Inclusion Criteria:

1. Study group Singleton pregnancies complicated with hypertension undergoing pre-labour CS at gestational age (34+0 to 40+0). These will be divided into 3 groups according to the type of disease either chronic hypertension (Group A), gestational hypertension (Group B) or preeclampsia (Group C).
2. Control group Singleton pregnancies undergoing elective pre-labour CS that are otherwise healthy.

Exclusion Criteria:

* Women with history of medical co-morbidities other than hypertension were excluded from the study. This includes the following: Renal diseases, autoimmune diseases, history of organ transplantation and immunosuppressive therapy, hematological diseases, history of thrombotic events, cardiopulmonary diseases, liver diseases, Acute and chronic inflammatory diseases.
* Pregnancy induced medical disorders like: Gestational thrombocytopenia.
* Multiple pregnancies.
* Abnormal placentation, i.e. Placenta previa and Morbidly adherent placenta.
* Fetal anomalies.
* vaginal deliveries and CS in labour.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosis of chronic hypertension, gestational hypertension and preeclampsia preeclampsia:Women with hypertension (>140/90 mmHg) and proteinuria (> 0.3 gm/day or ≥+1 by dipstick urine analysis at ≥ 20 weeks of gestation or protein-to-creatinine ratio of ≥ 0.30).
  Gestational hypertension: Women with systolic blood pressure is 140 mmHg or more or a diastolic blood pressure of 90 mmHg or more, or both, on two occasions at least 4 hours apart after 20 weeks of gestation, in a woman with a previously normal blood pressure.
  Chronic hypertension: It means systolic blood pressure of 140 mmHg or more, a diastolic blood pressure of 90 mmHg or more, or both, that is diagnosed or present before pregnancy or before 20 weeks of gestation on two occasions at least 4 hours apart.
  Patients are finally classified to PE with severe features, PE without severe features, Gestational hypertension, chronic hypertension and chronic hypertension with superimposed PE.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-20 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Telocytes in placenta and umbilical cord | Immediately after delivery of the placenta during cesarian section of pregnancies with gestational age (34-40) weeks
  The number and distribution of Telocytes by immunohistochemistry in placenta and umbilical cord vessels wall.

SECONDARY OUTCOMES:
Telocytes Morphology in relation to disease severity | Immediately after delivery of the placenta during cesarian section of pregnancies with gestational age (34-40) weeks
  Characterization of telocyte morphology using electron microscopy, comparing umbilical artery indices in different groups and its correlation to abundance of telocytes in examined tissues.

CONTACTS AND LOCATIONS:
Locations (1):
- Hatem Awaga, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided